CLINICAL TRIAL: NCT04873713
Title: Effects of Magnetic Tape Over Internal Hip Rotation in Patients With Low Back Pain
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Logistics and infrastructure problems
Sponsor: Francisco Selva (Other)
Responsible Party: Sponsor-Investigator, Francisco Selva, Principal Investigator, Clínica Dr. Francisco Selva
Organization: Clínica Dr. Francisco Selva (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12409331
Record Dates: First submitted 2021-04-26; First posted 2021-05-05 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Low Back Pain
Keywords: hip rotation; Magnetic tape; Kinovea® program; range of motion
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No Intervention: internal hip rotation (No Intervention): internal hip rotation pre measurement with knee and hip flexion at 90º, internal hip rotation will be performed
- Experimental: internal hip rotation (Experimental): internal hip rotation post experimental application measurement with Magnetic tape Application with knee and hip flexion at 90º, internal hip rotation will be performed
  Interventions: Device: Magnetic Tape® aplicación
- Placebo Comparator: internal hip rotation (Placebo Comparator): internal hip rotation post placebo application measurement with Placebo tape Application with knee and hip flexion at 90o, internal hip rotation will be performed
  Interventions: Device: Kinesiology Tape

INTERVENTIONS:
Device: Magnetic Tape® aplicación — Magnetic tape® is applied without creating any tension over low back
  Arms: Experimental: internal hip rotation
Device: Kinesiology Tape — Kinesiology Tape is applied without creating any tension over low back
  Arms: Placebo Comparator: internal hip rotation

SUMMARY:
The tape will be applied on the lumbar area bilateralemten to the spine without creating any tension.

The possible variation in the range of motion in internal hip rotation is measured with the KInovea program. A kinesiology tape was used as a placebo tape and the magnetic tape was used in a randomized experimental way.

DETAILED DESCRIPTION:
A triple-blind cross-sectional observational study is designed where subjects with low back pain will be selected and blinded to receive the Magnetic Tape® (tape with magnetic effects of less than 2 Gauss) or placebo Tape. Likewise, the evaluator who puts the Magnetic Tape® does not know what material he is using, as it is supplied by another researcher. The patient does not know what tape will be placed on him.

The recommendations of the "Consolidated Standards of Reporting Trials" (CONSORT) will be followed. All participants will receive a participant information sheet and sign informed consent. Patients aged 18 to 65 years with low back pain will be recruited from different private clinics in the city of Valencia, Spain.

The hypothesis is that when Magnetic Tape® comes into contact with electromagnetic fields such as those generated by living beings, due to the movement of electrical charges (ions), as defined by Ampere's Law, the domains of the tape are oriented or aligned in parallel with the external magnetic field creating a magnetic flux with a north pole and a south pole. This generated field in turn produces a magnetic induction proportional to the variation of the magnetic flux, as defined by the Faraday Law.

This electric potential produces a redistribution of the electric charge (ions) generating a magnetic field due to the orientation of the tape domains, then exerting a force on the moving charges within the electrolyte.

Physiological, Lorentz's Law, regulating Magnetic Tape® aberrant electromagnetic fields.

The protocol for data collection will be as follows:

After signing the informed consent and data protection, the groups with low back pain will be formed that will receive the application of both Magnetic Tape® and the intervention of a placebo tape. To avoid that the order of the intervention influences the results of the study, the subjects will be randomized into two different groups, Group A and Group B. Group A will receive Magnetic tape® and Group B will do the opposite. The next day the other tape will be applied Passive joint ROM of both hips is assessed by placing the patient in a supine position with 90º hip and knee flexion, performing passive internal hip rotation. The video camera is located perpendicular (ceiling) to the ipsilateral knee and hip to make recordings and measurements.

The tapes will be placed on the paravertebral skin from L1 to L5 without creating tension.

Subsequently, both hips are assessed again, performing passive internal hip rotation again and recording the degrees of range of motion.

Each subject will be your control since one day a tape will be placed and the next day the other.

Neither application has to be painful.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with low back pain.
* Subjects aged 18-65 years.

Exclusion Criteria:

* Tape allergies
* Adhesive allergies
* Pregnant
* People with pacemakers
* People who have any contraindication of electromagnetic fields
* People with neurological diseases
* Taking any medication that may interact with magnetic fields.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-07-04 (Estimated); Primary Completion 2021-07-04 (Estimated); Study Completion 2021-07-04 (Estimated)

PRIMARY OUTCOMES:
Range of motion | Changes from Range of motion first assessment before placing the tapes and inmediatly after placing experimental tape and placebo tape.
  Maximum degrees of internal hip rotation measured with the Kinovea® program. Validated Video Program

CONTACTS AND LOCATIONS:
Locations (1):
- Clínica Dr. Francisco Selva (Fisioterapia), Valencia, Spain

IPD SHARING:
Plan to Share IPD: No